CLINICAL TRIAL: NCT02045589
Title: A Phase I, Multicenter, Open-label, Dose Escalation Study of Intratumoral Injections of VCN-01 Oncolytic Adenovirus With Intravenous Gemcitabine and Abraxane® in Advanced Pancreatic Cancer
Brief Title: A Phase I Dose Escalation Study of Intratumoral VCN-01 Injections With Gemcitabine and Abraxane® in Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theriva Biologics SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-VCNA-002; 2012-005556-42 (EudraCT Number)
Record Dates: First submitted 2014-01-21; First posted 2014-01-27 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Pancreatic Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma
Keywords: Cancer; Pancreatic adenocarcinoma; Locally advanced; Metastatic; Gemcitabine; Oncolytic virus; Abraxane®
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation, Combination (Experimental): Three intratumoral administrations of VCN-01 oncolytic adenovirus every 28 days in combination with Abraxane® and Gemcitabine.
  Interventions: Genetic: VCN-01; Drug: Gemcitabine; Drug: Abraxane®

INTERVENTIONS:
Genetic: VCN-01 — Genetically modified human adenovirus encoding human PH20 hyaluronidase
Drug: Gemcitabine — 1000 mg/m2 intravenous administration
Drug: Abraxane® — 125 mg/m2 intravenous administration

SUMMARY:
The purpose of this study is to determine the safety and tolerability of three intratumoral injections of VCN-01 combined with Abraxane®/gemcitabine, and to determine the recommended phase II dose of VCN-01 combined with Abraxane®/gemcitabine.

DETAILED DESCRIPTION:
Investigational treatment is a dose-escalation regimen consisting of three VCN-01 intratumoral injections (once every 28 days at the same dose) in combination with intravenous Abraxane® and gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female patients aged 18 years or over
* Patients must provide written informed consent
* Life expectancy above 3 months
* Patients willing to comply with treatment follow-up, and to accept a biopsy at day 29 after initiation of the treatment
* Patients with histologically confirmed diagnosis of unresectable pancreatic adenocarcinoma with symptoms related to the primary tumor. Abraxane® plus Gemcitabine should be the appropriate standard of care to be administered.
* ECOG Performance status 0 or 1
* Adequate baseline organ function (hematologic, liver, renal and nutritional)
* Use a reliable method of contraception in fertile men and women

Exclusion Criteria:

* Active infection or other serious illness or autoimmune disease
* Treatment with live attenuated vaccines in the last three weeks
* Known chronic liver disease (liver cirrhosis, chronic hepatitis)
* Treatment with another investigational agent within its five half-lives prior to VCN-01 infusion
* Viral syndrome diagnosed during the two weeks before inclusion
* Chronic immunosuppressive therapy
* Known concurrent malignant hematologic or solid disease
* Pregnancy or lactation. Patients must agree to use effective contraception or be surgically sterile.
* Patients receiving full-dose anticoagulant / antiplatelet therapy
* Patients with Li Fraumeni syndrome or with previous known retinoblastoma protein pathway germinal deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability by means of Adverse Events (AEs) and laboratory data | At least 6 months
Recommended Phase 2 Dose (RP2D) of VCN-01 in combination with Gemcitabine and Abraxane® by determination of highest feasible dose (MFD) and any Dose Limiting Toxicities | At least 6 months

SECONDARY OUTCOMES:
Presence of VCN-01 in tumor | Day 21-28
  Determination of VCN-01 viral genome copies in tumor biopsy
Viral Pharmacokinetics | 48 h
  Determination of VCN-01 half-life by analyzing viral genome copies in blood
Viral Shedding | Up to day 71
  At least up to 6 months follow-up in patients at the Maximum Tolerated Dose (MTD)
Neutralizing antibodies anti-VCN-01 | 30 days after end of treatment phase
  At least up to 6 months follow-up in patients at the MTD
Preliminary anti-tumor activity by Overall Response Rate (ORR) | CT or MRI scans every 8 weeks until disease progression
Preliminary anti-tumor activity by Progression Free Survival (PFS) | CT or MRI scans every 8 weeks until disease progression

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

REFERENCES:
- [Derived] Bazan-Peregrino M, Garcia-Carbonero R, Laquente B, Alvarez R, Mato-Berciano A, Gimenez-Alejandre M, Morgado S, Rodriguez-Garcia A, Maliandi MV, Riesco MC, Moreno R, Ginesta MM, Perez-Carreras M, Gornals JB, Prados S, Perea S, Capella G, Alemany R, Salazar R, Blasi E, Blasco C, Cascallo M, Hidalgo M. VCN-01 disrupts pancreatic cancer stroma and exerts antitumor effects. J Immunother Cancer. 2021 Nov;9(11):e003254. doi: 10.1136/jitc-2021-003254. PMID 35149591